CLINICAL TRIAL: NCT00050271
Title: An Open-Label, Dose-Escalation Pilot Study of Acetyl-L-Carnitine for the Treatment of Dideoxynucleoside-Associated Distal Symmetric Peripheral Neuropathy
Brief Title: Acetyl-L-Carnitine for the Treatment of NRTI-Associated Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Neurologic AIDS Research Consortium (NARC) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5157; 10004 (Registry Identifier: DAIDS ES); ACTG A5157
Record Dates: First submitted 2002-12-03; First posted 2002-12-04 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Peripheral Nervous System Diseases
Keywords: Acetylcarnitine; Dideoxynucleosides; Epidermis; Biopsy; Immunohistochemistry; Nerve Fibers; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases | interventions — Acetylcarnitine

INTERVENTIONS:
Drug: Acetyl-L-carnitine

SUMMARY:
The purpose of this study is to determine if acetyl-L-carnitine (ALC) reduces pain, numbness, and tingling in the feet and legs of patients with nucleoside reverse transcriptase inhibitor (NRTI)-associated peripheral neuropathy. Another purpose is to determine if ALC is safe and tolerable in HIV patients who have taken certain anti-HIV drugs.

DETAILED DESCRIPTION:
Distal symmetric peripheral neuropathy (DSPN) is the most frequent neurologic complication of HIV infection and its treatments. NRTIs, particularly dideoxy-NRTIs, represent a significant risk factor for developing neuropathy. To date, there are no effective treatments for DSPN. Studies of nonneuronal tissues indicate a beneficial effect of ALC in HIV-1 seropositive individuals, but the role of ALC levels in patients with DSPN is unclear. Despite conflicting data, carnitine and its derivatives are still commonly used.

Patients will have a screening visit and visits at entry and Weeks 6, 12, 18, and 24. Patients are required to fast (no food or drink except water) for 4-12 hours for the screening visit, entry visit, and at Weeks 12 and 24. Targeted physical examinations, blood chemistries, liver function tests, HIV-1 RNA, CD4/CD8 cell counts, hematology, and lactate assessments will be done. Patients will also have a small skin biopsy at entry and Week 24. Patients will begin with 1 tablet of ALC twice daily and escalate dosage to a target dose of 3 tablets daily. They will remain on the 3-tablet dose or a maximum tolerated dose for the duration of the study (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Viral load <= 10,000 copies/ml within 60 days of entry
* On stable antiretroviral medication for 8 weeks prior to entry and plan on staying on current regimen for the duration of the study
* Currently taking at least one dideoxynucleoside analogue. Patients discontinuing their dideoxynucleoside analogues or changing their antiretroviral regimen after entry will remain on study drug and continue with the study requirements and evaluation visits.
* No significant systemic antiretroviral toxicity
* Evidence of predominantly sensory neuropathy, as determined from an examination by a neurologist
* Ongoing neuropathy of any duration
* Negative pregnancy test performed at screening and within 24 hours of study entry
* Agree not to become pregnant or to impregnate; agree to use acceptable methods of contraception

Exclusion Criteria:

* ALC or similar drug within 90 days of entry
* Active AIDS-defining opportunistic infection (OI) or OI-defining condition within 30 days prior to entry
* Any condition or history of any condition, other than that related to HIV infection or antiretroviral therapy, that would add confusion to the diagnosis of dideoxynucleoside analogue-associated DSPN
* Pregnancy or breast-feeding
* Active malignancy
* Seizure disorder or history of seizure within 90 days of entry
* Current or history of bipolar disorder
* Certain drugs within 30 days of study entry
* Addition of certain pain medication during the 60 days prior to study entry
* Allergy/sensitivity to study drug or its formulations
* Any condition that, in the opinion of the site investigator, would interfere with the study requirements
* Myelopathy
* Use of investigational agents that are not FDA-approved within 30 days of study entry, except when approved by the study chair. Investigational antiretroviral drugs available through expanded access or through AACTG trials will be allowed if they do not conflict with study criteria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Valcour, M.D., Study Chair — University of Hawaii; Russell Bartt, M.D., Study Chair — Cook County Hospital and Rush-Presbyterian St. Luke's Medical Center
Locations (11):
- United States (10):
  - Stanford CRS, Palo Alto, California
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Wulff EA, Wang AK, Simpson DM. HIV-associated peripheral neuropathy: epidemiology, pathophysiology and treatment. Drugs. 2000 Jun;59(6):1251-60. doi: 10.2165/00003495-200059060-00005. PMID 10882161
- [Background] Simpson DM, Katzenstein D, Haidich B, Millington D, Yiannoutsos C, Schifitto G, McArthur J; AIDS Clinical Trials Group Protocol 291/860 Study Team. Plasma carnitine in HIV-associated neuropathy. AIDS. 2001 Nov 9;15(16):2207-8. doi: 10.1097/00002030-200111090-00025. No abstract available. PMID 11684949
- [Background] Polydefkis M, Yiannoutsos CT, Cohen BA, Hollander H, Schifitto G, Clifford DB, Simpson DM, Katzenstein D, Shriver S, Hauer P, Brown A, Haidich AB, Moo L, McArthur JC. Reduced intraepidermal nerve fiber density in HIV-associated sensory neuropathy. Neurology. 2002 Jan 8;58(1):115-9. doi: 10.1212/wnl.58.1.115. PMID 11781415
- [Background] Scarpini E, Sacilotto G, Baron P, Cusini M, Scarlato G. Effect of acetyl-L-carnitine in the treatment of painful peripheral neuropathies in HIV+ patients. J Peripher Nerv Syst. 1997;2(3):250-2. PMID 10975731